CLINICAL TRIAL: NCT05466240
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging Trial to Evaluate Pharmacokinetics, Pharmacodynamics, and Safety of AT-752 in Patients With Dengue Infection
Brief Title: Study of AT-752 in Patients With Dengue Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to deprioritize the dengue program
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-02A-002
Record Dates: First submitted 2022-06-21; First posted 2022-07-20 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Dengue Fever
Keywords: Dengue; Vector borne disease; Infections; Virus disease; Viral; RNA virus; Hemorrhagic fevers
MeSH Terms: conditions — Dengue; Vector Borne Diseases; Infections; Virus Diseases; Hemorrhagic Fevers, Viral | interventions — AT-752

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Eligible subjects will be randomized to receive either AT-752 or matching placebo orally 3 times a day (TID) for 5 days in Cohort 1 of the study.
  Subsequent cohorts will receive AT-752/placebo either twice a day (BID) or TID
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AT-752 750-mg TID for 5 days (Active Comparator): Tablet; 750-mg, Three (3) times a day for 5-days
  Interventions: Drug: AT-752; Drug: Placebo
- AT-752 Dose A for 5 days (Active Comparator): Tablet; Dose A, for 5-days
  Interventions: Drug: AT-752; Drug: Placebo
- AT-752 Dose B for 5 days (Active Comparator): Tablet; Dose B, for 5-days
  Interventions: Drug: AT-752; Drug: Placebo

INTERVENTIONS:
Drug: AT-752 — AT-752 for 5 days
Drug: Placebo — Placebo for 5 days

SUMMARY:
The Phase 2 study will be conducted in adult patients with confirmed Dengue infection and will investigate safety, PK, and pharmacodynamics (PD) in this population. The study will be conducted in several dosing cohorts to enable dose selection for subsequent trials

ELIGIBILITY:
Key Inclusion Criteria:

* 18-55 years of age at time of screening
* Fever ≥38°C (or feeling feverish) with onset during the previous 48 hours
* Live/work in or recent travel to dengue endemic area
* Positive test confirming Dengue (DENV) on a NS1 antigen test or reverse transcription-polymerase chain reaction (RT-PCR) assay
* Negative rapid diagnostic test result for Coronavirus (SARS-CoV-2) and Influenza A and B

Key Exclusion Criteria:

* Pregnant, plans to become pregnant within 90 days of screening, or breast feeding.
* Has previously received any investigational or approved vaccine for dengue
* Previous history of HIV, chronic hepatitis B infection, or current hepatitis C infection (from medical history)
* Use of any antiviral drug within 30 days or within 5 half-lives of the active drug or metabolite (for long-acting antivirals)
* Current use of anticoagulant or antiplatelet drugs or documented medical history of bleeding disorders
* Current use of medications for treatment of inflammatory bowel disease or documented medical history of chronic gastrointestinal disease including inflammatory bowel disease
* Immunocompromised due to use of immunosuppressive drugs including systemic corticosteroids (inhaled or topical corticosteroids are allowed) or any current disease or condition
* Evidence of severe dengue disease
* Confirmed or suspected Coronavirus (SARS-CoV-2) infection or contact with patients with confirmed SARS-CoV2 infection within 7 days prior to screening
* Other clinically significant medical conditions or laboratory abnormalities, as described in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- Brazil (11):
  - Atea Study Site, Belo Horizonte
  - Atea Study Site, Campo Grande
  - Atea Study Site, Cuiabá
  - Atea Study Site, Manaus
  - Atea Study Site, Natal
  - Atea Study Site, Porto Velho
  - Atea Study Site, Recife
  - Atea Study Site, Ribeirão Preto
  - Atea Study Site, Rio de Janeiro
  - Atea Study Site, São José do Rio Preto
  - Atea Study Site, São Paulo
- Colombia (5):
  - Atea Study Site, Aguazul
  - Atea Study Site, Antioquia
  - Atea Study Site, Cali
  - Atea Study Site, Girardot
  - Atea Study Site, Yopal
- Atea Study Site, Machala, Ecuador
- India (4):
  - Atea Study Site, Guwahati
  - Atea Study Site, Kanpur
  - Atea Study Site, Lucknow
  - Atea Study Site, Sūrat
- Malaysia (2):
  - Atea Study Site, Kuala Terengganu
  - Atea Study Site, Perai
- Peru (2):
  - Atea Study Site, Ica
  - Atea Study Site, Iquitos
- Philippines (3):
  - Atea Study Site, Iloilo City
  - Atea Study Site, Las Piñas
  - Atea Study Site, Quezon City
- Atea Study Site, Kaohsiung City, Taiwan
- Thailand (2):
  - Atea Study Site, Bangkok
  - Atea Study Site, Khon Kaen
- Atea Study Site, Hanoi, Vietnam

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo TID for 5 Days: Tablet; Placebo, Three (3) times a day for 5-days
  Placebo: Placebo for 5 days
Period: Overall Study
Arm/Group | AT-752 750-mg TID for 5 Days | Placebo TID for 5 Days
Started | 14 | 7
Completed | 12 | 7
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AT-752 750-mg TID for 5 Days | Placebo TID for 5 Days | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 7 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (8.53) | 28.0 (5.54) | 30.1 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Philippines | 2 | 2 | 4
  Thailand | 5 | 2 | 7
  India | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Dengue (DENV) Viral Load From Baseline
Description: To investigate the antiviral activity of AT-752 versus placebo in terms of reduction of DENV RNA from baseline in adult subjects with confirmed DENV infection
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 14, Day 28
Population: Number of subjects with available viral load for baseline and the particular post-baseline timepoint.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | AT-752 750-mg TID for 5 Days | Placebo TID for 5 Days
Number analyzed (Participants) | 13 | 7
log10 copies/mL
  Baseline Viral Load: number analyzed (Participants) | 12 | 7
  Baseline Viral Load | 5.8 (2.0) | 4.6 (2.5)
  Day 2: number analyzed (Participants) | 12 | 7
  Day 2 | -1.3 (1.1) | -0.8 (0.9)
  Day 3: number analyzed (Participants) | 9 | 6
  Day 3 | -2.8 (1.3) | -1.2 (1.3)
  Day 4: number analyzed (Participants) | 11 | 7
  Day 4 | -3.3 (1.8) | -1.2 (1.7)
  Day 5: number analyzed (Participants) | 11 | 7
  Day 5 | -3.3 (1.8) | -1.8 (2.6)
  Day 6: number analyzed (Participants) | 11 | 7
  Day 6 | -3.3 (1.8) | -1.9 (2.5)
  Day 8: number analyzed (Participants) | 11 | 7
  Day 8 | -3.4 (1.8) | -1.9 (2.5)
  Day 14: number analyzed (Participants) | 11 | 7
  Day 14 | -3.3 (1.9) | -1.9 (2.5)
  Day 28: number analyzed (Participants) | 11 | 7
  Day 28 | -3.4 (1.8) | -1.9 (2.5)
Statistical Analysis 1: Comparison: AT-752 750-mg TID for 5 Days vs Placebo TID for 5 Days; Test type: Equivalence — For each post-baseline collection time point, treatment difference and p-value comparing the mean change in viral load from baseline between treatment arms from an analysis of covariance model with covariate baseline viral load; p < 0.95, ANCOVA

2. Secondary Outcome: Pharmacokinetic (PK) Endpoint
Description: Maximum plasma concentration (Cmax) of AT-281
Time Frame: Day 3: 0, 0.5, 1, 2, 4, 6 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AT-752 750-mg TID for 5 Days
Number analyzed (Participants) | 11
ng/mL | 2390 (2460)

3. Secondary Outcome: Pharmacokinetic (PK) Endpoint
Description: Area under the concentration-time curve (AUCtau) of AT-281
Time Frame: Day 3: 0, 0.5, 1, 2, 4, 6 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | AT-752 750-mg TID for 5 Days
Number analyzed (Participants) | 11
h*ng/mL | 4270 (2750)

ADVERSE EVENTS:
Time Frame: Day 28
Arm/Group | AT-752 750-mg TID for 5 Days | Placebo TID for 5 Days
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/7
Other Adverse Events (participants affected / at risk) | 10/14 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT-752 750-mg TID for 5 Days (N=14) | Placebo TID for 5 Days (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AT-752 750-mg TID for 5 Days (N=14) | Placebo TID for 5 Days (N=7)
Vomiting (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Fatigue (General disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Hematocrit increased (Investigations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early discontinuation leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may publish or present results pertaining to the PI's activities after the first publication of the multicentre clinical trial results. Publications must be submitted for review by Sponsor before submission. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (3):
  • Study Protocol: Original Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT05466240/Prot_000.pdf
  • Study Protocol: Amendment 1 (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT05466240/Prot_001.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT05466240/SAP_002.pdf